CLINICAL TRIAL: NCT02912871
Title: A Pilot Clinical Trial of the Feasibility, Safety and Efficacy of Subthalamotomy Using the ExAblate Transcranial System to Treat the Cardinal Motor Features of Parkinson's Disease
Brief Title: Subthalamotomy by ExAblate Transcranial System to Treat Motor Features of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: Insightech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD003E
Record Dates: First submitted 2016-08-19; First posted 2016-09-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson's Disease
Keywords: subthalamotomy; motor features; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- MRIgHIFU unilateral subthalamotomy (Experimental): Unilateral Subthalamotomy performed by MRI guided High intensity focused ultrasound in a single session.
  Interventions: Other: MRIgHIFU unilateral subthalamotomy

INTERVENTIONS:
Other: MRIgHIFU unilateral subthalamotomy — High Intensity focused ultrasound unilateral subthalamotomy: Unilateral thermolesion in the Subthalamic nucleus performed by High Intensity Focused ultrasound

SUMMARY:
Based on published animal and human studies, ExAblate Transcranial subthalamotomy can be as safe and as effective as any of the surgical treatments within the currently accepted standard of care including radiofrequency lesioning and Deep Brain Stimulation (DBS). A unilateral lesion of the subthalamic nucleus has shown reduction of contralateral motor symptoms in Parkinson's disease (PD). Using ExAblate Transcranial Magnetic Resonance guided High Intensity Focused Ultrasound (MRgHIFU) to create the subthalamotomy has several potential advantages over current therapies including the fact that transcranial lesioning can be performed in a precise manner with simultaneous as well as continuous clinical and radiographic monitoring. If the potential of ExAblate Transcranial subthalamotomy can be realized, it could supplant radiofrequency and radiosurgery techniques and provide a viable alternative procedure for subjects considering DBS.

DETAILED DESCRIPTION:
This ExAblate Transcranial system was built atop the ExAblate Body system technology, which has received EMA and CE approvals for the treatment of uterine fibroids and bone metastasis palliation, and is currently being evaluated under various EMA Investigational Device Exemptions "IDE". It should be noted that the ExAblate Transcranial/Neuro has received CE approval (Dec-2012).

There are many potential advantages for applying ExAblate Transcranial subthalamotomy for the treatment of idiopathic PD:

* The procedure is transcranial, requiring no incision, no burr hole, and no electrode. The risk of hemorrhagic complication should be reduced, and this procedure should eliminate the risk of infectious complications.
* Unlike stereotactic radiosurgery, ExAblate Transcranial system does not use ionizing radiation and does not carry a risk of radiation-induced tumorigenesis. The effects are immediate and not latent as with radiosurgery.
* Unlike radiofrequency ablation, ExAblate Transcranial system thermal lesioning can be performed without open surgery.
* The ExAblate treatment can be monitored in real-time with MRI and MR-thermal feedback which permits immediate confirmation of the targeting process. Additionally, the treatment can be monitored with clinical testing.
* Unlike DBS treatment, there is no implanted hardware, no concern of interference with external sources of electromagnetic noise, no need for extensive follow-up for programming, and no need for periodic battery replacement.

ExAblate Transcranial treatments may represent a simpler treatment algorithm for a patient suffering from a complicated disease process like PD. Hours of clinic time will be saved from DBS device management and replacement and health care costs may be greatly reduced.

- Rational for ExAblate Transcranial System subthalamotomy for the Treatment of PD Conceptually, lesioning the subthalamus seems logical since preclinical studies have confirmed the role of the subthalamic nucleus in the development of parkinsonism and by the fact that the experimental Parkinsonian state by MPTP can be relieved by exocytotic or thermolytic lesions of the STN. Furthermore, clinical studies of deep brain stimulation targeting the subthalamic nucleus have proven that this nucleus is the most effective for the treatment of advanced Parkinson's disease.

From a clinical perspective, unilateral subthalamotomy for medication-refractory Parkinson's disease certainly has proven beneficial in the alleviation of contralateral off-medication motor symptoms in several series. The largest and best reported experience comes from the CIREN (La Habana, Cuba) where this project was initiated and directed by Prof. Jose Obeso over a 10 years period leading to a large accumulated experience. This was described for 89 patients followed for up to 36 months. In these reports, significant improvements were noted on UPDRS ratings with bradykinesia, rigidity and tremor. Improvements remained at two years and were most pronounced for tremor. With regards to the "on" state, contralateral dyskinesia was reduced during the two-year study and the mean dose of Levodopa was decreased by 34-47% while the total on time without dyskinesia increased fourfold. In the study significant reductions in part three of the off-medication UPDRS were noted at 12 (50%), 24 (30%), and 36 months (18%) following unilateral subthalamotomy. In the "on" state, contralateral dyskinesia improved throughout the 3-year study period although ipsilateral dyskinesia progressively worsened during this time. In a limited number of patients bilateral staged ( N-7) and simultaneous ( N-11) subthalamotomy was carried out without major adverse effects and highly significant motor improvement. Cognitive changes were specifically ascertained prospectively without evidence of deterioration. More recently, the impact of unilateral subthalamotomy on inhibitory mechanisms was also reported from the same study group. Unexpectedly, speed of stopping an initiated action was improved after STN lesion.

Subthalamotomy has never been widely accepted because of concerns for hemiballismus primarily due to observations in humans with stroke in the region of the subthalamus (Purdon Martin 1927) and by the confirmation in the 1940's by Whittier and Mettler who were able to experimentally reproduce this by subthalamic lesions in primates. Arguments against such dogma were amply discussed years ago leading to the understanding that the parkinsonian state modifies the threshold to hemiballism after STN lesion.

The ExAblate modality permits a very precise focused lesion to be created without disruption of other motor pathways or nuclei. In order to test the feasibility of using the ExAblate Neuro system for the ablation of the subthalamic nucleus two patients (University of Virginia) were active-sham treated using a sublethal dose of energy (50-54⁰C). The subjects were observed for 30 days without developing any adverse effects like worsening involuntary movements. Since there were no adverse effects of worsening involuntary movements, the actual second stage treatment was then performed. Again, no adverse effects of worsening involuntary movements were observed. The safety profile remains favorable.

Interestingly, the rationale for choosing target temperatures of 50-54⁰C as a ' subtherapeutic/test' lesion was based on the experience acquired during the feasibility study for Essential Tremor under IDE # G10016969 and preclinical lesioning in a swine model. In 15 patients with ET, the typical onset of neurologic phenomena (ie sensory symptoms) or tremor suppression is observed when the peak voxel temperatures on MR thermography reached the low 50's ⁰C. It was observed that the tremor effect first occurs during the titrated lesioning process with transient suppression of postural and rest tremor. Later at higher temperatures of 55-65⁰C, the tremor effect becomes more lasting. Also T2 signal change on MRI is not typically visible acutely in human thalamus until peak voxel temperatures approach this 55-65⁰C range. These higher temperatures resulted in thalamotomy volumes comparable to traditional radiofrequency lesions where the diameter became maximal at 1 week (mean=171 mm3) and measured 6.8mm in diameter. Soon by one and three months, HIFU thalamotomy volumes subsided to 55 and 14 mm3, respectively.

Thus, small lesions with reversible clinical effects would occurre by confining the first, subtherapeutic/test lesion to 50-54⁰C. The therapeutic treatment goal must be to perform the final, peak voxel temperatures of 55-65⁰C which will result in a substantial target ablation which is analogous to the volume achieved with contemporary RF lesioning.

The rationale for unilateral subthalamotomy for advanced PD is summarized as follows:

1. A well-placed stereotactic lesion is similarly efficacious to DBS.
2. Stereotactic radiofrequency subthalamotomy has been shown to ameliorate the motor features of PD .
3. The risk for involuntary movements like hemichorea-ballism following subthalamotomy in humans is about 15% but only in the 9% of patients a second procedure (pallidotomy) was needed to treat the dyskinesias.
4. Studies of DBS in PD have consistently shown equivalent results between the stereotactic targets: STN and GPi.
5. The subthalamus is amenable to an image-guided ablation because it is small and easily visualized with contemporary MRI.
6. DBS, while effective for advanced PD, has complexities for patients, their caregivers, and their doctors and potentially carries a higher risk than ExAblate mediated lesion.

Summary Based on published animal and human studies, ExAblate Transcranial subthalamotomy can be as safe and as effective as any of the surgical treatments within the currently accepted standard of care including RF lesioning and DBS. A unilateral lesion of the subthalamic nucleus has shown reduction of contralateral motor symptoms in PD. Using ExAblate Transcranial MRgHIFU to create the subthalamotomy has several potential advantages over current therapies including the fact that transcranial lesioning can be performed in a precise manner with simultaneous as well as continuous clinical and radiographic monitoring. If the potential of ExAblate Transcranial subthalamotomy can be realized, it could supplant radiofrequency and radiosurgery techniques and provide a viable alternative procedure for subjects considering DBS.

This study will include ten Parkinson's disease patients who will be treated with unilateral subthalamotomy performed by MRIgHIFU and followed in an open-label fashion for up to 6 months to demonstrate safety and sustained benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subjects who are able and willing to give informed consent and able to attend all study visits through 6 Months
3. Subjects with a diagnosis of PD by United Kingdom Brain Bank Criteria as confirmed by a movement disorder neurologist at the site
4. Predominant disability from one side of the body (i.e unilateral or markedly asymmetric disease) as determined by a movement disorders neurologist
5. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry, if possible.
6. Topographic coordinates of the subthalamic nucleus are localizable on Magnetic resonance imaging (MRI) so that it can be targeted by the ExAblate device.
7. Subject is able to communicate sensations during the ExAblate Transcranial procedure.

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS).
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA) or Mattis Dementia Rating Scale of 120 or lower.
7. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
8. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory.
9. Legal incapacity or limited legal capacity as determined by the neuropsychologist
10. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) as manifested by one (or more) of the following occurring within the preceding 12-month period:

    * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
    * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
    * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
    * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
11. Subjects with unstable cardiac status including:

    * Unstable angina pectoris on medication
    * Subjects with documented myocardial infarction within six months of protocol entry
    * Significant congestive heart failure defined with ejection fraction < 40
    * Subjects with unstable ventricular arrhythmias
    * Subjects with atrial arrhythmias that are not rate-controlled
12. Severe hypertension (diastolic Blood Pressure > 100 on medication)
13. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy
14. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
15. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or international normalized ratio (INR) coagulation studies exceeding the institution's laboratory standard
16. Patient with severely impaired renal function with estimated glomerular filtration rate <30milliliter/minute/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis;
17. Subjects with standard contraindications for MRI imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
18. Significant claustrophobia that cannot be managed with mild medication.
19. Subject who weigh more than the upper weight limit of the MRI table and who cannot fit into the MRI scanner
20. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
21. History of intracranial hemorrhage
22. History of multiple strokes, or a stroke within past 6 months
23. Subjects with a history of seizures within the past year
24. Subjects with malignant brain tumors
25. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
26. Any illness that in the investigator's opinion preclude participation in this study.
27. Subjects unable to communicate with the investigator and staff.
28. Pregnancy or lactation.
29. Subjects who have an Overall Skull Density Ratio (SDR) of 0.3 (±0.05) or less as calculated from the screening Cranial Tomography scan (CT).

    * It should be noted that for those candidates whose SDR ratio score is within the standard deviation, full technical assessment should be performed and reviewed by study investigator with the support of the sponsor.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
All causes of morbidity | within the first 6 months (plus minus 1 month) after treatment
  Number of treatment-related adverse events as assessed by CTCAE v4.0
Efficacy | 6 months
  Improvement in the score of the Movement Disorders Unified Parkinson's Disease Rating Scale III (MDS-UPDRS III) that evaluates motor features of PD. The scale will be assessed pretreatment and after intervention and the reduction after treatment in the total MDS-UPDRS III score and the score in the treated hemibody will be measured. MDS-UPDRS III is a scale that assesses all the motor features of PD (akinesia, tremor, rigidity, gait disturbance). Score range between 0 (no presence of motor features) and 132 (maximum score for all items).

SECONDARY OUTCOMES:
MDS-UPDRS I | 6 months
  MDS-UPDRS I evaluates non-motor symptoms of PD. Scores of the scales will be measured pretreatment and after procedure and compared.
MDS-UPDRS II | 6 months
  MDS-UPDRS II evaluates dependence in daily life activities. Scores of the scales will be measured pretreatment and after procedure and compared.
MDS-UPDRS IV | 6 months
  MDS-UPDRS IV evaluates presence and impact of motor complications (i.e. motor fluctuations and dyskinesia).
  Scores of the scales will be measured pretreatment and after procedure and compared.
Dyskinesia severity as assessed through the Dyskinesia rating scale | 6 months
  Dyskinesia rating scale assesses the presence of involuntary movements
Levodopa equivalent medication usage (milligrams) when applicable | 6 months
Patient and Clinician Global Impression of Change | 6 months
Quality of life assessment with PDQ-39 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Obeso, MD, PhD, Principal Investigator — CINAC, HM Puerta del Sur. Avda. Carlos V nº 70. CP 28938. Móstoles MADRID (SPAIN) Tel: +34 91 2673201; Email: consulta.hmcinac@hmhospitales.com

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elias WJ, Huss D, Voss T, Loomba J, Khaled M, Zadicario E, Frysinger RC, Sperling SA, Wylie S, Monteith SJ, Druzgal J, Shah BB, Harrison M, Wintermark M. A pilot study of focused ultrasound thalamotomy for essential tremor. N Engl J Med. 2013 Aug 15;369(7):640-8. doi: 10.1056/NEJMoa1300962. PMID 23944301
- [Background] Lipsman N, Schwartz ML, Huang Y, Lee L, Sankar T, Chapman M, Hynynen K, Lozano AM. MR-guided focused ultrasound thalamotomy for essential tremor: a proof-of-concept study. Lancet Neurol. 2013 May;12(5):462-8. doi: 10.1016/S1474-4422(13)70048-6. Epub 2013 Mar 21. PMID 23523144
- [Background] Alvarez L, Macias R, Pavon N, Lopez G, Rodriguez-Oroz MC, Rodriguez R, Alvarez M, Pedroso I, Teijeiro J, Fernandez R, Casabona E, Salazar S, Maragoto C, Carballo M, Garcia I, Guridi J, Juncos JL, DeLong MR, Obeso JA. Therapeutic efficacy of unilateral subthalamotomy in Parkinson's disease: results in 89 patients followed for up to 36 months. J Neurol Neurosurg Psychiatry. 2009 Sep;80(9):979-85. doi: 10.1136/jnnp.2008.154948. Epub 2009 Feb 9. PMID 19204026
- [Derived] Martinez-Fernandez R, Natera-Villalba E, Manez Miro JU, Rodriguez-Rojas R, Marta Del Alamo M, Pineda-Pardo JA, Ammann C, Obeso I, Mata-Marin D, Hernandez-Fernandez F, Gasca-Salas C, Matarazzo M, Alonso-Frech F, Obeso JA. Prospective Long-term Follow-up of Focused Ultrasound Unilateral Subthalamotomy for Parkinson Disease. Neurology. 2023 Mar 28;100(13):e1395-e1405. doi: 10.1212/WNL.0000000000206771. Epub 2023 Jan 11. PMID 36631272
- [Derived] Rodriguez-Rojas R, Pineda-Pardo JA, Manez-Miro J, Sanchez-Turel A, Martinez-Fernandez R, Del Alamo M, DeLong M, Obeso JA. Functional Topography of the Human Subthalamic Nucleus: Relevance for Subthalamotomy in Parkinson's Disease. Mov Disord. 2022 Feb;37(2):279-290. doi: 10.1002/mds.28862. Epub 2021 Dec 3. PMID 34859498
- [Derived] Martinez-Fernandez R, Rodriguez-Rojas R, Del Alamo M, Hernandez-Fernandez F, Pineda-Pardo JA, Dileone M, Alonso-Frech F, Foffani G, Obeso I, Gasca-Salas C, de Luis-Pastor E, Vela L, Obeso JA. Focused ultrasound subthalamotomy in patients with asymmetric Parkinson's disease: a pilot study. Lancet Neurol. 2018 Jan;17(1):54-63. doi: 10.1016/S1474-4422(17)30403-9. Epub 2017 Dec 5. PMID 29203153